CLINICAL TRIAL: NCT06712251
Title: Early Feasibility Study of the Velocity™ Percutaneous Arterio-Venous Fistula System
Brief Title: Early Feasibility Study of the Velocity™ Percutaneous Arterio-Venous Fistula System for Creating Hemodialysis Vascular Access
Acronym: VENOS-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venova Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0687
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis; End Stage Renal Disease (ESRD)
Keywords: Dialysis Access; Hemodialysis; AV Fistula; Percutaneous AVF
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Velocity Percutaneous Arterio-Venous Fistula System (Experimental)
  Interventions: Device: Velocity pAVF System

INTERVENTIONS:
Device: Velocity pAVF System — The Velocity Percutaneous Arterio-Venous Fistula System consists of a percutaneous method designed to create an arteriovenous fistula for hemodialysis vascular access.
  Other Names: pAVF; endoAVF

SUMMARY:
The Velocity Percutaneous Arterio-Venous System is a minimally invasive method of creating hemodialysis vascular access. The study aims to understand clinical efficacy and initial clinical safety data of the device.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4/5 or ESRD
* Eligible for a native surgical proximal forearm radiocephalic arteriovenous fistula following assessment by the principal investigator and study sponsor
* Cubital perforating vein diameter ⩾ 2.0 and ⩽ 5.0 mm
* Proximal radial artery diameter ⩾ 2.0 and ⩽ 4.0 mm
* Willing and competent to give written informed consent
* Willing and able to complete all study assessments and follow-up requirements

Exclusion Criteria:

* Distance between Proximal Radial Artery and Cubital Perforating Vein > 3 mm
* Subject study extremity systolic blood pressure < 100mmHg Known central venous stenosis of > 50% ipsilateral to the study extremity
* Any obstruction of superficial venous outflow from intended device implant site to the axillary vein
* Subjects with occlusion of the ulnar or radial artery at any level or an abnormal Allen's test
* Any previous dialysis vascular access procedures in the study extremity
* History of access related hand ischemia from a previous hemodialysis vascular access of the non-study extremity which required intervention or access abandonment
* Upper extremity venous occlusion and/or vessel abnormality of the study extremity that precludes endovascular AVF creation as determined by principal investigator or study sponsor
* Evidence of active systemic infections on day of the procedure or infection at the procedure access site within the past 7 days
* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Any contraindication to antiplatelet therapy
* Currently being treated with another investigational device or drug
* Known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated
* Uncontrolled or poorly controlled diabetes defined as a HbA1C > 10%
* Known hypercoagulable condition, bleeding diathesis or coagulation disorder
* Receiving anti-coagulant therapy that cannot be safely held in the peri-procedural period
* Edema of the study extremity
* Scheduled kidney transplant within 6 months of enrollment
* Peripheral white blood cell count < 1,500 cells/microL or > 13,000 cells/microL and neutrophil > 80%
* Platelet count < 75,000 cells/ microL
* Serum procalcitonin level > 0.75 ng/mL for subjects with central venous catheters
* Current diagnosis of carcinoma (unless in remission > 1 year)
* Pregnant or currently breast feeding
* History of substance abuse or anticipated to be non- compliant with medical care or study requirements based on investigator judgment
* Allergies to nickel or nickel titanium alloy (NiTi) or any of the components of the Velocity Implant or Delivery System
* Any other medical condition that in the opinion of the investigator would put the welfare of the subject at risk or confound interpretation of the study data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Physiologic Maturation | 6 weeks
  The proportion of participants that reach the binary outcome of Physiologic Maturation (mature/unmature). Physiologic Maturation is a composite measure, reached when Duplex ultrasound demonstrates a brachial artery blood flow of ≥ 500 ml/min and an outflow vein diameter of ≥ 5 mm.
Serious Adverse Device Effect | 30 days
  Any Serious Adverse Event that reasonably suggests is caused by the device or procedure

SECONDARY OUTCOMES:
Functional Maturation | 3 months
  The number of participants with successful two needle cannulation for 75% of dialysis sessions over a consecutive 4 weeks period following pAVF creation
Unassisted Functional Maturation | 3 months
  The number of participants that reach functional maturation without any endovascular or surgical interventions to the pAVF to facilitate maturation and/or manage complications
Time to First Hemodialysis | Up to 52 weeks
  The interval from the time of pAVF creation to the first hemodialysis session using 2-needles in the ESRD subgroup
Number of Catheter Days | Up to 52 weeks
  The number of days from pAVF creation to central venous catheter removal in the ESRD subgroup.
Total Reinterventions | 12 months
  All reinterventions related to the access will be captured over the life of the access until abandonment or when the subject exits the study.
Freedom from Reintervention | Up to 104 weeks
  The duration from the time of access creation until the first occurrence of a reintervention required to maintain or restore patency of the pAVF
Technical Success | Day of study intervention
  Intraprocedural duplex ultrasound demonstrating arterialized flow in the cephalic vein
Primary Patency | 6 months
  The time of access creation until the first occurrence of any reintervention to maintain or reestablish patency or until access abandonment
Primary Assisted Patency | 6 months
  The time from access creation to the first reintervention to maintain patency, including reinterventions intended to prevent thrombosis or restenosis, without the occurrence of thrombosis or abandonment of the access
Cumulative Patency | 6 months
  The interval from the time of access creation or intervention until the final abandonment of the access, inclusive of all successful interventions to maintain or restore patency
Freedom from Serious Adverse Events | Up to 104 weeks
  The time from access creation to the first occurrence of any serious adverse event (SAE)
Functional Patency | 12 months
  Elapsed time from functional maturation to abandonment of the access site

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Trinity Research Group, Dothan, Alabama
  - Apex Research, Riverside, California
  - American Access Care of Jacksonville, Jacksonville, Florida
  - Texas Research Institute, Fort Worth, Texas
  - STAR Vascular, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF